CLINICAL TRIAL: NCT03768414
Title: A Phase III Randomized Trial of Gemcitabine, Cisplatin, and Nab-Paclitaxel Versus Gemcitabine and Cisplatin in Newly Diagnosed, Advanced Biliary Tract Cancers
Brief Title: Gemcitabine Hydrochloride and Cisplatin With or Without Nab-Paclitaxel in Treating Patients With Newly Diagnosed Advanced Biliary Tract Cancers
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: SWOG Cancer Research Network (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: S1815; NCI-2018-01920 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); S1815 (Other: SWOG); S1815 (Other: CTEP); U10CA180888 (NIH)
Record Dates: First submitted 2018-12-06; First posted 2018-12-07 (Actual); Results first posted 2024-10-22 (Actual); Last update posted 2026-01-12 (Actual); Status verified 2026-01

CONDITIONS: Stage III Distal Bile Duct Cancer AJCC v8; Stage III Gallbladder Cancer AJCC v8; Stage III Intrahepatic Cholangiocarcinoma AJCC v8; Stage IIIA Distal Bile Duct Cancer AJCC v8; Stage IIIA Gallbladder Cancer AJCC v8; Stage IIIA Intrahepatic Cholangiocarcinoma AJCC v8; Stage IIIB Distal Bile Duct Cancer AJCC v8; Stage IIIB Gallbladder Cancer AJCC v8; Stage IIIB Intrahepatic Cholangiocarcinoma AJCC v8; Stage IV Distal Bile Duct Cancer AJCC v8; Stage IV Gallbladder Cancer AJCC v8; Stage IV Intrahepatic Cholangiocarcinoma AJCC v8; Stage IVA Gallbladder Cancer AJCC v8; Stage IVB Gallbladder Cancer AJCC v8; Unresectable Extrahepatic Bile Duct Carcinoma; Unresectable Gallbladder Carcinoma; Unresectable Intrahepatic Cholangiocarcinoma
MeSH Terms: conditions — Gallbladder Neoplasms; Cholangiocarcinoma | interventions — Cisplatin; 1,2-diaminocyclohexaneplatinum II citrate; Platinum; Gemcitabine; 130-nm albumin-bound paclitaxel; Albumin-Bound Paclitaxel; Taxes

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Arm I (nab-paclitaxel, cisplatin, gemcitabine hydrochloride) (Experimental): Patients receive nab-paclitaxel IV over 30 minutes, cisplatin IV over 60 minutes, and gemcitabine hydrochloride IV over 30 minutes on days 1 and 8. Courses repeat every 21 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Cisplatin; Drug: Gemcitabine Hydrochloride; Drug: Nab-paclitaxel
- Arm II (cisplatin, gemcitabine hydrochloride) (Experimental): Patients receive cisplatin IV over 60 minutes and gemcitabine hydrochloride IV over 30 minutes on days 1 and 8. Courses repeat every 21 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Cisplatin; Drug: Gemcitabine Hydrochloride

INTERVENTIONS:
Drug: Cisplatin — Given IV
  Other Names: Abiplatin; Blastolem; Briplatin; CDDP; Cis-diammine-dichloroplatinum; Cis-diamminedichloridoplatinum; Cis-diamminedichloro Platinum (II); Cis-diamminedichloroplatinum; Cis-dichloroammine Platinum (II); Cis-platinous Diamine Dichloride; Cis-platinum; Cis-platinum II; Cis-platinum II Diamine Dichloride; Cismaplat; Cisplatina; Cisplatinum; Cisplatyl; Citoplatino; Citosin; Cysplatyna; DDP; Lederplatin; Metaplatin; Neoplatin; Peyrone's Chloride; Peyrone's Salt; Placis; Plastistil; Platamine; Platiblastin; Platiblastin-S; Platinex; Platinol; Platinol- AQ; Platinol-AQ; Platinol-AQ VHA Plus; Platinoxan; Platinum; Platinum Diamminodichloride; Platiran; Platistin; Platosin
Drug: Gemcitabine Hydrochloride — Given IV
  Other Names: dFdCyd; Difluorodeoxycytidine Hydrochloride; Gemzar; LY-188011; LY188011
Drug: Nab-paclitaxel — Given IV
  Other Names: ABI 007; ABI-007; Abraxane; Albumin-bound Paclitaxel; Albumin-Stabilized Nanoparticle Paclitaxel; Nanoparticle Albumin-bound Paclitaxel; Nanoparticle Paclitaxel; paclitaxel albumin-stabilized nanoparticle formulation; Protein-bound Paclitaxel
  Arms: Arm I (nab-paclitaxel, cisplatin, gemcitabine hydrochloride)

SUMMARY:
This phase III trial studies how well gemcitabine hydrochloride and cisplatin given with or without nab-paclitaxel work in treating patients with newly diagnosed biliary tract cancers that have spread to other places in the body. Drugs used in chemotherapy, such as gemcitabine hydrochloride, cisplatin, and nab-paclitaxel, work in different ways to stop the growth of tumor cells, either by killing the cells, by stopping them from dividing, or by stopping them from spreading. It is not known if giving gemcitabine hydrochloride and cisplatin with or without nab-paclitaxel may work better at treating biliary tract cancers.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To compare overall survival (OS) in patients with untreated, advanced biliary cancers treated with gemcitabine hydrochloride (gemcitabine) and cisplatin (GC) versus those treated with gemcitabine, cisplatin, and nab-Paclitaxel (GCN).

SECONDARY OBJECTIVES:

I. To compare progression-free survival (PFS) in patients treated with GC versus GCN.

II. To compare overall response rate (ORR), complete and partial, confirmed and unconfirmed, in the subset of patients with measurable disease treated with GC versus GCN.

III. To compare disease control rate (confirmed and unconfirmed; complete response + partial response + stable disease) (DCR) in patients treated with GC versus GCN.

IV. To evaluate the frequency and severity of toxicity associated with GC and GCN in the patient population.

V. To explore the correlation between change in cancer antigen 19-9 (CA19-9) levels from baseline to post-treatment (after 3 cycles) and overall response rate, in each treatment arm separately and in the total cohort.

ADDITIONAL OBJECTIVES:

I. To bank tissue and blood for future translational medicine studies.

OUTLINE: Patients are randomized to 1 of 2 arms.

ARM I: Patients receive nab-paclitaxel intravenously (IV) over 30 minutes, cisplatin IV over 60 minutes, and gemcitabine hydrochloride IV over 30 minutes on days 1 and 8. Courses repeat every 21 days in the absence of disease progression or unacceptable toxicity.

ARM II: Patients receive cisplatin IV over 60 minutes and gemcitabine hydrochloride IV over 30 minutes on days 1 and 8. Courses repeat every 21 days in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up every 6 months for 2 years and then at the end of year 3.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have histologically or cytologically confirmed intrahepatic cholangiocarcinoma, extrahepatic cholangiocarcinoma, or gallbladder cancer

  * NOTE: Pathology report must be uploaded in Rave. Histology report must be consistent with an adenocarcinoma with pancreaticobiliary primary assuming there are no pancreatic lesions and other primaries are ruled out per local standard
* Patients must have documented metastatic or locally advanced unresectable disease on computed tomography (CT) or magnetic resonance (MR) imaging CT scans or MRIs used to assess measurable disease. Must have been completed within 28 days prior to registration. CT scans or MRIs used to assess non-measurable disease must have been completed within 42 days prior to registration. All disease must be assessed and documented on the Baseline Tumor Assessment Form
* Patient must not have a current diagnosis of ampullary cancer
* Patients must not have received prior systemic therapy for the current metastatic or locally advanced biliary cancer
* Patient must not have received adjuvant therapy within 6 months prior to registration
* Patients must have a complete medical history and physical exam within 28 days prior to registration
* Patients must have a Zubrod performance status of 0 or 1
* Patients must not have a history of peripheral neuropathy of grade 2 or greater by Common Terminology Criteria for Adverse Events (CTCAE) 5.0. In CTCAE version 5.0 grade 2 sensory neuropathy is defined as ?moderate symptoms; limiting instrumental activities of daily living (ADLs)?
* Absolute neutrophil count (ANC) >= 1,500/mcL (obtained within 28 days prior to registration)
* Platelets >= 100,000/mcL (obtained within 28 days prior to registration)
* Hemoglobin >= 8 g/dL (obtained within 28 days prior to registration)
* Serum albumin >= 2.8 g/dL (obtained within 28 days prior to registration)
* Total bilirubin =< 1.5 x institutional upper limit of normal (IULN) (except patients with Gilbert?s syndrome, who must have a direct bilirubin < 1.5 mg/dL) (obtained within 28 days prior to registration)
* Serum glutamic-oxaloacetic transaminase (SGOT) (aspartate aminotransferase [AST]) and serum glutamate pyruvate transaminase (SGPT) (alanine aminotransferase [ALT]) =< 8 x IULN (obtained within 28 days prior to registration)
* Serum creatinine =< IULN OR calculated creatinine clearance >= 60 mL/min (obtained within 28 days prior to registration)
* Patients must have CA19-9 obtained within 42 days prior to registration
* Patients must have sodium, potassium, bicarbonate, chloride, blood urea nitrogen (BUN), calcium, total protein, magnesium, and alkaline phosphatase obtained within 28 days prior to registration
* Patients must not have an active infection requiring systemic therapy
* No other prior malignancy is allowed except for the following: adequately treated basal cell or squamous cell skin cancer, in situ cervical cancer, adequately treated stage I or II cancer from which the patient is currently in complete remission, or any other cancer from which the patient has been disease free for two years
* Patients must not be pregnant or nursing. Women/men of reproductive potential must have agreed to use an effective contraceptive method. A woman is considered to be of "reproductive potential" if she has had menses at any time in the preceding 12 consecutive months. In addition to routine contraceptive methods, "effective contraception" also includes heterosexual celibacy and surgery intended to prevent pregnancy (or with a side-effect of pregnancy prevention) defined as a hysterectomy, bilateral oophorectomy or bilateral tubal ligation. However, if at any point a previously celibate patient chooses to become heterosexually active during the time period for use of contraceptive measures outlined in the protocol, he/she is responsible for beginning contraceptive measures
* Sites must seek additional patient consent for the future use of specimens
* Patients must be informed of the investigational nature of this study and must sign and give written informed consent in accordance with institutional and federal guidelines
* As a part of the Oncology Patient Enrollment Network (OPEN) registration process the treating institution's identity is provided in order to ensure that the current (within 365 days) date of institutional review board approval for this study has been entered in the system

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 452 (Actual)
Dates: Start 2019-02-07 (Actual); Primary Completion 2023-10-04 (Actual); Study Completion 2024-10-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Rachna Shroff, Principal Investigator — SWOG Cancer Research Network
Locations (692):
- United States (692):
  - Anchorage Associates in Radiation Medicine, Anchorage, Alaska
  - Anchorage Radiation Therapy Center, Anchorage, Alaska
  - Alaska Breast Care and Surgery LLC, Anchorage, Alaska
  - Alaska Oncology and Hematology LLC, Anchorage, Alaska
  - Alaska Women's Cancer Care, Anchorage, Alaska
  - Anchorage Oncology Centre, Anchorage, Alaska
  - Katmai Oncology Group, Anchorage, Alaska
  - Providence Alaska Medical Center, Anchorage, Alaska
  - CTCA at Western Regional Medical Center, Goodyear, Arizona
  - Kingman Regional Medical Center, Kingman, Arizona
  - Cancer Center at Saint Joseph's, Phoenix, Arizona
  - Mayo Clinic Hospital in Arizona, Phoenix, Arizona
  - Mayo Clinic in Arizona, Scottsdale, Arizona
  - University of Arizona Cancer Center-Orange Grove Campus, Tucson, Arizona
  - Banner University Medical Center - Tucson, Tucson, Arizona
  - University of Arizona Cancer Center-North Campus, Tucson, Arizona
  - Mercy Hospital Fort Smith, Fort Smith, Arkansas
  - CHI Saint Vincent Cancer Center Hot Springs, Hot Springs, Arkansas
  - Baptist Memorial Hospital and Fowler Family Cancer Center - Jonesboro, Jonesboro, Arkansas
  - University of Arkansas for Medical Sciences, Little Rock, Arkansas
  - Mission Hope Medical Oncology - Arroyo Grande, Arroyo Grande, California
  - PCR Oncology, Arroyo Grande, California
  - Providence Saint Joseph Medical Center/Disney Family Cancer Center, Burbank, California
  - Community Cancer Institute, Clovis, California
  - University Oncology Associates, Clovis, California
  - City of Hope Corona, Corona, California
  - City of Hope Comprehensive Cancer Center, Duarte, California
  - Los Angeles County-USC Medical Center, Los Angeles, California
  - USC / Norris Comprehensive Cancer Center, Los Angeles, California
  - Fremont - Rideout Cancer Center, Marysville, California
  - City of Hope Mission Hills, Mission Hills, California
  - USC Norris Oncology/Hematology-Newport Beach, Newport Beach, California
  - UC Irvine Health/Chao Family Comprehensive Cancer Center, Orange, California
  - Stanford Cancer Institute Palo Alto, Palo Alto, California
  - University of California Davis Comprehensive Cancer Center, Sacramento, California
  - Salinas Valley Memorial, Salinas, California
  - UCSF Medical Center-Mission Bay, San Francisco, California
  - Pacific Central Coast Health Center-San Luis Obispo, San Luis Obispo, California
  - City of Hope - Santa Clarita, Santa Clarita, California
  - Mission Hope Medical Oncology - Santa Maria, Santa Maria, California
  - City of Hope South Pasadena, South Pasadena, California
  - Gene Upshaw Memorial Tahoe Forest Cancer Center, Truckee, California
  - City of Hope Upland, Upland, California
  - City of Hope West Covina, West Covina, California
  - Rocky Mountain Regional VA Medical Center, Aurora, Colorado
  - Penrose-Saint Francis Healthcare, Colorado Springs, Colorado
  - Rocky Mountain Cancer Centers-Penrose, Colorado Springs, Colorado
  - Porter Adventist Hospital, Denver, Colorado
  - Mercy Medical Center, Durango, Colorado
  - Southwest Oncology PC, Durango, Colorado
  - Mountain Blue Cancer Care Center, Golden, Colorado
  - Rocky Mountain Cancer Centers-Lakewood, Lakewood, Colorado
  - Saint Anthony Hospital, Lakewood, Colorado
  - Littleton Adventist Hospital, Littleton, Colorado
  - Longmont United Hospital, Longmont, Colorado
  - Rocky Mountain Cancer Centers-Longmont, Longmont, Colorado
  - Parker Adventist Hospital, Parker, Colorado
  - Rocky Mountain Cancer Centers-Parker, Parker, Colorado
  - Saint Mary Corwin Medical Center, Pueblo, Colorado
  - Rocky Mountain Cancer Centers - Pueblo, Pueblo, Colorado
  - Rocky Mountain Cancer Centers-Thornton, Thornton, Colorado
  - Smilow Cancer Hospital-Derby Care Center, Derby, Connecticut
  - Smilow Cancer Hospital Care Center-Fairfield, Fairfield, Connecticut
  - Smilow Cancer Hospital Care Center - Guiford, Guilford, Connecticut
  - Smilow Cancer Hospital Care Center at Saint Francis, Hartford, Connecticut
  - Smilow Cancer Center/Yale-New Haven Hospital, New Haven, Connecticut
  - Yale University, New Haven, Connecticut
  - Yale-New Haven Hospital North Haven Medical Center, North Haven, Connecticut
  - Smilow Cancer Hospital-Orange Care Center, Orange, Connecticut
  - Smilow Cancer Hospital-Torrington Care Center, Torrington, Connecticut
  - Smilow Cancer Hospital Care Center-Trumbull, Trumbull, Connecticut
  - Smilow Cancer Hospital-Waterbury Care Center, Waterbury, Connecticut
  - Smilow Cancer Hospital Care Center - Waterford, Waterford, Connecticut
  - Beebe South Coastal Health Campus, Frankford, Delaware
  - Beebe Medical Center, Lewes, Delaware
  - Delaware Clinical and Laboratory Physicians PA, Newark, Delaware
  - Helen F Graham Cancer Center, Newark, Delaware
  - Medical Oncology Hematology Consultants PA, Newark, Delaware
  - Christiana Care Health System-Christiana Hospital, Newark, Delaware
  - Beebe Health Campus, Rehoboth Beach, Delaware
  - TidalHealth Nanticoke / Allen Cancer Center, Seaford, Delaware
  - Christiana Care Health System-Wilmington Hospital, Wilmington, Delaware
  - Sibley Memorial Hospital, Washington D.C., District of Columbia
  - AdventHealth Altamonte, Altamonte Springs, Florida
  - Mount Sinai Comprehensive Cancer Center at Aventura, Aventura, Florida
  - AdventHealth Celebration, Celebration, Florida
  - Regional Cancer Center-Lee Memorial Health System, Fort Myers, Florida
  - Mayo Clinic in Florida, Jacksonville, Florida
  - AdventHealth Kissimmee, Kissimmee, Florida
  - Mount Sinai Medical Center, Miami Beach, Florida
  - AdventHealth Medical Group Urology at Orlando, Orlando, Florida
  - AdventHealth Orlando, Orlando, Florida
  - AdventHealth East Orlando, Orlando, Florida
  - AdventHealth Winter Park, Winter Park, Florida
  - Hawaii Cancer Care Inc-POB II, Honolulu, Hawaii
  - Island Urology, Honolulu, Hawaii
  - Queen's Cancer Cenrer - POB I, Honolulu, Hawaii
  - Queen's Medical Center, Honolulu, Hawaii
  - Straub Clinic and Hospital, Honolulu, Hawaii
  - University of Hawaii Cancer Center, Honolulu, Hawaii
  - Hawaii Cancer Care Inc-Liliha, Honolulu, Hawaii
  - Kuakini Medical Center, Honolulu, Hawaii
  - Queen's Cancer Center - Kuakini, Honolulu, Hawaii
  - The Cancer Center of Hawaii-Liliha, Honolulu, Hawaii
  - Kapiolani Medical Center for Women and Children, Honolulu, Hawaii
  - Wilcox Memorial Hospital and Kauai Medical Clinic, Lihue, Hawaii
  - Hawaii Cancer Care - Savio, ‘Aiea, Hawaii
  - Pali Momi Medical Center, ‘Aiea, Hawaii
  - Queen's Cancer Center - Pearlridge, ‘Aiea, Hawaii
  - The Cancer Center of Hawaii-Pali Momi, ‘Aiea, Hawaii
  - Saint Alphonsus Cancer Care Center-Boise, Boise, Idaho
  - Saint Luke's Mountain States Tumor Institute, Boise, Idaho
  - Saint Alphonsus Cancer Care Center-Caldwell, Caldwell, Idaho
  - Kootenai Medical Center, Coeur d'Alene, Idaho
  - Walter Knox Memorial Hospital, Emmett, Idaho
  - Saint Luke's Cancer Institute - Fruitland, Fruitland, Idaho
  - Idaho Urologic Institute-Meridian, Meridian, Idaho
  - Saint Luke's Cancer Institute - Meridian, Meridian, Idaho
  - Saint Alphonsus Medical Center-Nampa, Nampa, Idaho
  - Saint Luke's Cancer Institute - Nampa, Nampa, Idaho
  - Kootenai Cancer Center, Post Falls, Idaho
  - Kootenai Cancer Clinic, Sandpoint, Idaho
  - Saint Luke's Cancer Institute - Twin Falls, Twin Falls, Idaho
  - Rush - Copley Medical Center, Aurora, Illinois
  - Illinois CancerCare-Bloomington, Bloomington, Illinois
  - Illinois CancerCare-Canton, Canton, Illinois
  - Memorial Hospital of Carbondale, Carbondale, Illinois
  - SIH Cancer Institute, Carterville, Illinois
  - Illinois CancerCare-Carthage, Carthage, Illinois
  - Centralia Oncology Clinic, Centralia, Illinois
  - Northwestern University, Chicago, Illinois
  - University of Illinois, Chicago, Illinois
  - Carle on Vermilion, Danville, Illinois
  - Cancer Care Specialists of Illinois - Decatur, Decatur, Illinois
  - Decatur Memorial Hospital, Decatur, Illinois
  - Northwestern Medicine Cancer Center Kishwaukee, DeKalb, Illinois
  - Illinois CancerCare-Dixon, Dixon, Illinois
  - Carle Physician Group-Effingham, Effingham, Illinois
  - Crossroads Cancer Center, Effingham, Illinois
  - Illinois CancerCare-Eureka, Eureka, Illinois
  - Illinois CancerCare-Galesburg, Galesburg, Illinois
  - Western Illinois Cancer Treatment Center, Galesburg, Illinois
  - Northwestern Medicine Cancer Center Delnor, Geneva, Illinois
  - Joliet Oncology-Hematology Associates Limited, Joliet, Illinois
  - Illinois CancerCare-Kewanee Clinic, Kewanee, Illinois
  - Northwestern Medicine Lake Forest Hospital, Lake Forest, Illinois
  - Illinois CancerCare-Macomb, Macomb, Illinois
  - Carle Physician Group-Mattoon/Charleston, Mattoon, Illinois
  - Good Samaritan Regional Health Center, Mount Vernon, Illinois
  - Cancer Care Center of O'Fallon, O'Fallon, Illinois
  - Illinois CancerCare-Ottawa Clinic, Ottawa, Illinois
  - Illinois CancerCare-Pekin, Pekin, Illinois
  - OSF Saint Francis Radiation Oncology at Pekin Cancer Treatment Center, Pekin, Illinois
  - Illinois CancerCare-Peoria, Peoria, Illinois
  - OSF Saint Francis Radiation Oncology at Peoria Cancer Center, Peoria, Illinois
  - Methodist Medical Center of Illinois, Peoria, Illinois
  - OSF Saint Francis Medical Center, Peoria, Illinois
  - Illinois CancerCare-Peru, Peru, Illinois
  - Valley Radiation Oncology, Peru, Illinois
  - Illinois CancerCare-Princeton, Princeton, Illinois
  - Genesis Cancer Center - Silvis, Silvis, Illinois
  - Southern Illinois University School of Medicine, Springfield, Illinois
  - Springfield Clinic, Springfield, Illinois
  - Memorial Medical Center, Springfield, Illinois
  - Southwest Illinois Health Services LLP, Swansea, Illinois
  - Carle Cancer Center, Urbana, Illinois
  - The Carle Foundation Hospital, Urbana, Illinois
  - Northwestern Medicine Cancer Center Warrenville, Warrenville, Illinois
  - Rush-Copley Healthcare Center, Yorkville, Illinois
  - IU Health North Hospital, Carmel, Indiana
  - Indiana University/Melvin and Bren Simon Cancer Center, Indianapolis, Indiana
  - Franciscan Health Indianapolis, Indianapolis, Indiana
  - Franciscan Saint Elizabeth Health - Lafayette East, Lafayette, Indiana
  - Woodland Cancer Care Center, Michigan City, Indiana
  - Franciscan Health Mooresville, Mooresville, Indiana
  - Reid Health, Richmond, Indiana
  - Union Hospital, Terre Haute, Indiana
  - Mary Greeley Medical Center, Ames, Iowa
  - McFarland Clinic PC - Ames, Ames, Iowa
  - McFarland Clinic PC-Boone, Boone, Iowa
  - Medical Oncology and Hematology Associates-West Des Moines, Clive, Iowa
  - Mercy Cancer Center-West Lakes, Clive, Iowa
  - Alegent Health Mercy Hospital, Council Bluffs, Iowa
  - Greater Regional Medical Center, Creston, Iowa
  - Genesis Medical Center - East Campus, Davenport, Iowa
  - Genesis Cancer Care Institute, Davenport, Iowa
  - Iowa Cancer Specialists, Davenport, Iowa
  - Iowa Methodist Medical Center, Des Moines, Iowa
  - Medical Oncology and Hematology Associates-Des Moines, Des Moines, Iowa
  - Broadlawns Medical Center, Des Moines, Iowa
  - Medical Oncology and Hematology Associates-Laurel, Des Moines, Iowa
  - Mercy Medical Center - Des Moines, Des Moines, Iowa
  - Iowa Lutheran Hospital, Des Moines, Iowa
  - McFarland Clinic PC-Trinity Cancer Center, Fort Dodge, Iowa
  - Trinity Regional Medical Center, Fort Dodge, Iowa
  - McFarland Clinic PC-Jefferson, Jefferson, Iowa
  - McFarland Clinic PC-Marshalltown, Marshalltown, Iowa
  - Siouxland Regional Cancer Center, Sioux City, Iowa
  - Methodist West Hospital, West Des Moines, Iowa
  - Mercy Medical Center-West Lakes, West Des Moines, Iowa
  - Lawrence Memorial Hospital, Lawrence, Kansas
  - Cancer Center of Kansas-Wichita Medical Arts Tower, Wichita, Kansas
  - Cancer Center of Kansas - Wichita, Wichita, Kansas
  - Flaget Memorial Hospital, Bardstown, Kentucky
  - Commonwealth Cancer Center-Corbin, Corbin, Kentucky
  - Saint Joseph Radiation Oncology Resource Center, Lexington, Kentucky
  - Saint Joseph Hospital East, Lexington, Kentucky
  - Saint Joseph London, London, Kentucky
  - Jewish Hospital, Louisville, Kentucky
  - The James Graham Brown Cancer Center at University of Louisville, Louisville, Kentucky
  - Saints Mary and Elizabeth Hospital, Louisville, Kentucky
  - Jewish Hospital Medical Center Northeast, Louisville, Kentucky
  - Jewish Hospital Medical Center South, Shepherdsville, Kentucky
  - LSU Health Baton Rouge-North Clinic, Baton Rouge, Louisiana
  - Louisiana Hematology Oncology Associates LLC, Baton Rouge, Louisiana
  - Mary Bird Perkins Cancer Center, Baton Rouge, Louisiana
  - Our Lady of the Lake Physicians Group - Medical Oncology, Baton Rouge, Louisiana
  - Medical Center of Baton Rouge, Baton Rouge, Louisiana
  - Ochsner High Grove, Baton Rouge, Louisiana
  - Louisiana State University Health Science Center, New Orleans, Louisiana
  - Ochsner Medical Center Jefferson, New Orleans, Louisiana
  - Harold Alfond Center for Cancer Care, Augusta, Maine
  - Eastern Maine Medical Center, Bangor, Maine
  - Waldo County General Hospital, Belfast, Maine
  - MaineHealth/SMHC Cancer Care and Blood Disorders-Biddeford, Biddeford, Maine
  - Lafayette Family Cancer Center-EMMC, Brewer, Maine
  - Stephens Memorial Hospital, Norway, Maine
  - Penobscot Bay Medical Center, Rockport, Maine
  - MaineHealth/SMHC Cancer Care and Blood Disorders-Sanford, Sanford, Maine
  - Maine Medical Partners - South Portland, South Portland, Maine
  - Johns Hopkins University/Sidney Kimmel Cancer Center, Baltimore, Maryland
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - Lowell General Hospital, Lowell, Massachusetts
  - UMass Memorial Medical Center - University Campus, Worcester, Massachusetts
  - University of Michigan Comprehensive Cancer Center, Ann Arbor, Michigan
  - Bronson Battle Creek, Battle Creek, Michigan
  - McLaren Cancer Institute-Bay City, Bay City, Michigan
  - Henry Ford Cancer Institute-Downriver, Brownstown, Michigan
  - McLaren Cancer Institute-Clarkston, Clarkston, Michigan
  - Henry Ford Macomb Hospital-Clinton Township, Clinton Township, Michigan
  - Henry Ford Medical Center-Fairlane, Dearborn, Michigan
  - Wayne State University/Karmanos Cancer Institute, Detroit, Michigan
  - Henry Ford Hospital, Detroit, Michigan
  - Weisberg Cancer Treatment Center, Farmington Hills, Michigan
  - McLaren Cancer Institute-Flint, Flint, Michigan
  - Singh and Arora Hematology Oncology PC, Flint, Michigan
  - Helen DeVos Children's Hospital at Spectrum Health, Grand Rapids, Michigan
  - Mercy Health Saint Mary's, Grand Rapids, Michigan
  - Spectrum Health at Butterworth Campus, Grand Rapids, Michigan
  - Allegiance Health, Jackson, Michigan
  - Bronson Methodist Hospital, Kalamazoo, Michigan
  - West Michigan Cancer Center, Kalamazoo, Michigan
  - Borgess Medical Center, Kalamazoo, Michigan
  - McLaren-Greater Lansing, Lansing, Michigan
  - Mid-Michigan Physicians-Lansing, Lansing, Michigan
  - McLaren Cancer Institute-Lapeer Region, Lapeer, Michigan
  - McLaren Cancer Institute-Macomb, Mount Clemens, Michigan
  - McLaren Cancer Institute-Central Michigan, Mount Pleasant, Michigan
  - Mercy Health Mercy Campus, Muskegon, Michigan
  - Lakeland Hospital Niles, Niles, Michigan
  - Cancer and Hematology Centers of Western Michigan - Norton Shores, Norton Shores, Michigan
  - Ascension Providence Hospitals - Novi, Novi, Michigan
  - Henry Ford Medical Center-Columbus, Novi, Michigan
  - Huron Medical Center PC, Port Huron, Michigan
  - Lake Huron Medical Center, Port Huron, Michigan
  - McLaren-Port Huron, Port Huron, Michigan
  - Spectrum Health Reed City Hospital, Reed City, Michigan
  - Lakeland Medical Center Saint Joseph, Saint Joseph, Michigan
  - Marie Yeager Cancer Center, Saint Joseph, Michigan
  - Henry Ford Macomb Health Center - Shelby Township, Shelby, Michigan
  - Ascension Providence Hospitals - Southfield, Southfield, Michigan
  - Munson Medical Center, Traverse City, Michigan
  - Henry Ford West Bloomfield Hospital, West Bloomfield, Michigan
  - Metro Health Hospital, Wyoming, Michigan
  - Riverwood Healthcare Center, Aitkin, Minnesota
  - Sanford Joe Lueken Cancer Center, Bemidji, Minnesota
  - Essentia Health Saint Joseph's Medical Center, Brainerd, Minnesota
  - Fairview Ridges Hospital, Burnsville, Minnesota
  - Minnesota Oncology - Burnsville, Burnsville, Minnesota
  - Cambridge Medical Center, Cambridge, Minnesota
  - Mercy Hospital, Coon Rapids, Minnesota
  - Essentia Health - Deer River Clinic, Deer River, Minnesota
  - Essentia Health Saint Mary's - Detroit Lakes Clinic, Detroit Lakes, Minnesota
  - Essentia Health Cancer Center, Duluth, Minnesota
  - Essentia Health Saint Mary's Medical Center, Duluth, Minnesota
  - Miller-Dwan Hospital, Duluth, Minnesota
  - Fairview Southdale Hospital, Edina, Minnesota
  - Lake Region Healthcare Corporation-Cancer Care, Fergus Falls, Minnesota
  - Essentia Health - Fosston, Fosston, Minnesota
  - Unity Hospital, Fridley, Minnesota
  - Essentia Health Hibbing Clinic, Hibbing, Minnesota
  - Fairview Clinics and Surgery Center Maple Grove, Maple Grove, Minnesota
  - Minnesota Oncology Hematology PA-Maplewood, Maplewood, Minnesota
  - Saint John's Hospital - Healtheast, Maplewood, Minnesota
  - Abbott-Northwestern Hospital, Minneapolis, Minnesota
  - Hennepin County Medical Center, Minneapolis, Minnesota
  - Health Partners Inc, Minneapolis, Minnesota
  - Monticello Cancer Center, Monticello, Minnesota
  - New Ulm Medical Center, New Ulm, Minnesota
  - Essentia Health - Park Rapids, Park Rapids, Minnesota
  - Fairview Northland Medical Center, Princeton, Minnesota
  - North Memorial Medical Health Center, Robbinsdale, Minnesota
  - Mayo Clinic in Rochester, Rochester, Minnesota
  - Park Nicollet Clinic - Saint Louis Park, Saint Louis Park, Minnesota
  - Regions Hospital, Saint Paul, Minnesota
  - United Hospital, Saint Paul, Minnesota
  - Essentia Health Sandstone, Sandstone, Minnesota
  - Saint Francis Regional Medical Center, Shakopee, Minnesota
  - Lakeview Hospital, Stillwater, Minnesota
  - Sanford Thief River Falls Medical Center, Thief River Falls, Minnesota
  - Essentia Health Virginia Clinic, Virginia, Minnesota
  - Ridgeview Medical Center, Waconia, Minnesota
  - Rice Memorial Hospital, Willmar, Minnesota
  - Minnesota Oncology Hematology PA-Woodbury, Woodbury, Minnesota
  - Sanford Cancer Center Worthington, Worthington, Minnesota
  - Fairview Lakes Medical Center, Wyoming, Minnesota
  - Baptist Memorial Hospital and Cancer Center-Golden Triangle, Columbus, Mississippi
  - The West Clinic - Corinth, Corinth, Mississippi
  - Baptist Cancer Center-Grenada, Grenada, Mississippi
  - Gulfport Memorial Hospital, Gulfport, Mississippi
  - Baptist Memorial Hospital and Cancer Center-Union County, New Albany, Mississippi
  - Baptist Memorial Hospital and Cancer Center-Oxford, Oxford, Mississippi
  - The West Clinic - Southaven, Southaven, Mississippi
  - Baptist Memorial Hospital and Cancer Center-Desoto, Southhaven, Mississippi
  - Saint Louis Cancer and Breast Institute-Ballwin, Ballwin, Missouri
  - Parkland Health Center-Bonne Terre, Bonne Terre, Missouri
  - Cox Cancer Center Branson, Branson, Missouri
  - Saint Francis Medical Center, Cape Girardeau, Missouri
  - Southeast Cancer Center, Cape Girardeau, Missouri
  - Saint Luke's Hospital, Chesterfield, Missouri
  - Siteman Cancer Center at Saint Peters Hospital, City of Saint Peters, Missouri
  - Siteman Cancer Center at West County Hospital, Creve Coeur, Missouri
  - Parkland Health Center - Farmington, Farmington, Missouri
  - Capital Region Southwest Campus, Jefferson City, Missouri
  - Freeman Health System, Joplin, Missouri
  - Mercy Hospital Joplin, Joplin, Missouri
  - Delbert Day Cancer Institute at PCRMC, Rolla, Missouri
  - Mercy Clinic-Rolla-Cancer and Hematology, Rolla, Missouri
  - Heartland Regional Medical Center, Saint Joseph, Missouri
  - Sainte Genevieve County Memorial Hospital, Sainte Genevieve, Missouri
  - Mercy Hospital Springfield, Springfield, Missouri
  - CoxHealth South Hospital, Springfield, Missouri
  - Saint Louis Cancer and Breast Institute-South City, St Louis, Missouri
  - Washington University School of Medicine, St Louis, Missouri
  - Mercy Hospital South, St Louis, Missouri
  - Siteman Cancer Center-South County, St Louis, Missouri
  - Missouri Baptist Medical Center, St Louis, Missouri
  - Siteman Cancer Center at Christian Hospital, St Louis, Missouri
  - Mercy Hospital Saint Louis, St Louis, Missouri
  - Missouri Baptist Sullivan Hospital, Sullivan, Missouri
  - Missouri Baptist Outpatient Center-Sunset Hills, Sunset Hills, Missouri
  - Mercy Hospital Washington, Washington, Missouri
  - Community Hospital of Anaconda, Anaconda, Montana
  - Billings Clinic Cancer Center, Billings, Montana
  - Bozeman Deaconess Hospital, Bozeman, Montana
  - Benefis Healthcare- Sletten Cancer Institute, Great Falls, Montana
  - Great Falls Clinic, Great Falls, Montana
  - Saint Peter's Community Hospital, Helena, Montana
  - Kalispell Regional Medical Center, Kalispell, Montana
  - Saint Patrick Hospital - Community Hospital, Missoula, Montana
  - Community Medical Hospital, Missoula, Montana
  - CHI Health Saint Francis, Grand Island, Nebraska
  - Heartland Hematology and Oncology, Kearney, Nebraska
  - CHI Health Good Samaritan, Kearney, Nebraska
  - Saint Elizabeth Regional Medical Center, Lincoln, Nebraska
  - Nebraska Methodist Hospital, Omaha, Nebraska
  - Alegent Health Immanuel Medical Center, Omaha, Nebraska
  - Hematology and Oncology Consultants PC, Omaha, Nebraska
  - Alegent Health Bergan Mercy Medical Center, Omaha, Nebraska
  - Alegent Health Lakeside Hospital, Omaha, Nebraska
  - Creighton University Medical Center, Omaha, Nebraska
  - Midlands Community Hospital, Papillion, Nebraska
  - Carson Tahoe Regional Medical Center, Carson City, Nevada
  - Cancer and Blood Specialists-Henderson, Henderson, Nevada
  - Comprehensive Cancer Centers of Nevada - Henderson, Henderson, Nevada
  - Comprehensive Cancer Centers of Nevada-Horizon Ridge, Henderson, Nevada
  - Las Vegas Cancer Center-Henderson, Henderson, Nevada
  - OptumCare Cancer Care at Seven Hills, Henderson, Nevada
  - 21st Century Oncology-Henderson, Henderson, Nevada
  - Comprehensive Cancer Centers of Nevada-Southeast Henderson, Henderson, Nevada
  - Las Vegas Urology - Green Valley, Henderson, Nevada
  - Las Vegas Urology - Pebble, Henderson, Nevada
  - Urology Specialists of Nevada - Green Valley, Henderson, Nevada
  - Las Vegas Urology - Pecos, Las Vegas, Nevada
  - Desert West Surgery, Las Vegas, Nevada
  - OptumCare Cancer Care at Oakey, Las Vegas, Nevada
  - University Medical Center of Southern Nevada, Las Vegas, Nevada
  - Hope Cancer Care of Nevada, Las Vegas, Nevada
  - Cancer and Blood Specialists-Shadow, Las Vegas, Nevada
  - Radiation Oncology Centers of Nevada Central, Las Vegas, Nevada
  - Urology Specialists of Nevada - Central, Las Vegas, Nevada
  - 21st Century Oncology, Las Vegas, Nevada
  - HealthCare Partners Medical Group Oncology/Hematology-Maryland Parkway, Las Vegas, Nevada
  - Sunrise Hospital and Medical Center, Las Vegas, Nevada
  - HealthCare Partners Medical Group Oncology/Hematology-San Martin, Las Vegas, Nevada
  - Las Vegas Prostate Cancer Center, Las Vegas, Nevada
  - Las Vegas Urology - Sunset, Las Vegas, Nevada
  - Radiation Oncology Centers of Nevada Southeast, Las Vegas, Nevada
  - 21st Century Oncology-Vegas Tenaya, Las Vegas, Nevada
  - Ann M Wierman MD LTD, Las Vegas, Nevada
  - Cancer and Blood Specialists-Tenaya, Las Vegas, Nevada
  - Comprehensive Cancer Centers of Nevada - Northwest, Las Vegas, Nevada
  - HealthCare Partners Medical Group Oncology/Hematology-Tenaya, Las Vegas, Nevada
  - Las Vegas Urology - Cathedral Rock, Las Vegas, Nevada
  - Las Vegas Urology - Smoke Ranch, Las Vegas, Nevada
  - OptumCare Cancer Care at MountainView, Las Vegas, Nevada
  - Urology Specialists of Nevada - Northwest, Las Vegas, Nevada
  - Alliance for Childhood Diseases/Cure 4 the Kids Foundation, Las Vegas, Nevada
  - Comprehensive Cancer Centers of Nevada - Town Center, Las Vegas, Nevada
  - Comprehensive Cancer Centers of Nevada-Summerlin, Las Vegas, Nevada
  - Summerlin Hospital Medical Center, Las Vegas, Nevada
  - Las Vegas Cancer Center-Medical Center, Las Vegas, Nevada
  - 21st Century Oncology-Fort Apache, Las Vegas, Nevada
  - Comprehensive Cancer Centers of Nevada, Las Vegas, Nevada
  - OptumCare Cancer Care at Fort Apache, Las Vegas, Nevada
  - Urology Specialists of Nevada - Southwest, Las Vegas, Nevada
  - HealthCare Partners Medical Group Oncology/Hematology-Centennial Hills, Las Vegas, Nevada
  - Comprehensive Cancer Centers of Nevada - Central Valley, Las Vegas, Nevada
  - University Cancer Center, Las Vegas, Nevada
  - Hope Cancer Care of Nevada-Pahrump, Pahrump, Nevada
  - Renown Regional Medical Center, Reno, Nevada
  - Saint Mary's Regional Medical Center, Reno, Nevada
  - Radiation Oncology Associates, Reno, Nevada
  - Dartmouth Hitchcock Medical Center, Lebanon, New Hampshire
  - Memorial Sloan Kettering Basking Ridge, Basking Ridge, New Jersey
  - Memorial Sloan Kettering Monmouth, Middletown, New Jersey
  - Memorial Sloan Kettering Bergen, Montvale, New Jersey
  - Rutgers Cancer Institute of New Jersey, New Brunswick, New Jersey
  - Holy Name Hospital, Teaneck, New Jersey
  - Lovelace Medical Center-Saint Joseph Square, Albuquerque, New Mexico
  - University of New Mexico Cancer Center, Albuquerque, New Mexico
  - New Mexico Oncology Hematology Consultants, Albuquerque, New Mexico
  - Presbyterian Kaseman Hospital, Albuquerque, New Mexico
  - Memorial Medical Center - Las Cruces, Las Cruces, New Mexico
  - Presbyterian Rust Medical Center/Jorgensen Cancer Center, Rio Rancho, New Mexico
  - Roswell Park Cancer Institute, Buffalo, New York
  - Memorial Sloan Kettering Commack, Commack, New York
  - Glens Falls Hospital, Glens Falls, New York
  - Memorial Sloan Kettering Westchester, Harrison, New York
  - Laura and Isaac Perlmutter Cancer Center at NYU Langone, New York, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - NYP/Weill Cornell Medical Center, New York, New York
  - University of Rochester, Rochester, New York
  - Stony Brook University Medical Center, Stony Brook, New York
  - James J Peters VA Medical Center, The Bronx, New York
  - Memorial Sloan Kettering Nassau, Uniondale, New York
  - Southeastern Medical Oncology Center-Clinton, Clinton, North Carolina
  - Southeastern Medical Oncology Center-Goldsboro, Goldsboro, North Carolina
  - Wayne Memorial Hospital, Goldsboro, North Carolina
  - Margaret R Pardee Memorial Hospital, Hendersonville, North Carolina
  - Onslow Memorial Hospital, Jacksonville, North Carolina
  - Southeastern Medical Oncology Center-Jacksonville, Jacksonville, North Carolina
  - Vidant Oncology-Kenansville, Kenansville, North Carolina
  - Vidant Oncology-Kinston, Kinston, North Carolina
  - Vidant Oncology-Richlands, Richlands, North Carolina
  - Sanford Bismarck Medical Center, Bismarck, North Dakota
  - Essentia Health Cancer Center-South University Clinic, Fargo, North Dakota
  - Sanford South University Medical Center, Fargo, North Dakota
  - Sanford Medical Center Fargo, Fargo, North Dakota
  - Sanford Broadway Medical Center, Fargo, North Dakota
  - Sanford Roger Maris Cancer Center, Fargo, North Dakota
  - Essentia Health - Jamestown Clinic, Jamestown, North Dakota
  - UHHS-Chagrin Highlands Medical Center, Beachwood, Ohio
  - Indu and Raj Soin Medical Center, Beavercreek, Ohio
  - Strecker Cancer Center-Belpre, Belpre, Ohio
  - Saint Elizabeth Boardman Hospital, Boardman, Ohio
  - Hematology and Oncology Associates Inc, Canton, Ohio
  - Mercy Medical Center, Canton, Ohio
  - Dayton Physicians LLC-Miami Valley South, Centerville, Ohio
  - Miami Valley Hospital South, Centerville, Ohio
  - Geauga Hospital, Chardon, Ohio
  - Adena Regional Medical Center, Chillicothe, Ohio
  - University of Cincinnati/Barrett Cancer Center, Cincinnati, Ohio
  - Good Samaritan Hospital - Cincinnati, Cincinnati, Ohio
  - Oncology Hematology Care Inc-Kenwood, Cincinnati, Ohio
  - Bethesda North Hospital, Cincinnati, Ohio
  - TriHealth Cancer Institute-Westside, Cincinnati, Ohio
  - TriHealth Cancer Institute-Anderson, Cincinnati, Ohio
  - Case Western Reserve University, Cleveland, Ohio
  - MetroHealth Medical Center, Cleveland, Ohio
  - Mount Carmel East Hospital, Columbus, Ohio
  - Columbus Oncology and Hematology Associates Inc, Columbus, Ohio
  - Riverside Methodist Hospital, Columbus, Ohio
  - Grant Medical Center, Columbus, Ohio
  - The Mark H Zangmeister Center, Columbus, Ohio
  - Mount Carmel Health Center West, Columbus, Ohio
  - Doctors Hospital, Columbus, Ohio
  - Good Samaritan Hospital - Dayton, Dayton, Ohio
  - Miami Valley Hospital, Dayton, Ohio
  - Dayton Physician LLC-Miami Valley Hospital North, Dayton, Ohio
  - Miami Valley Hospital North, Dayton, Ohio
  - Dayton Veterans Affairs Medical Center, Dayton, Ohio
  - Delaware Health Center-Grady Cancer Center, Delaware, Ohio
  - Grady Memorial Hospital, Delaware, Ohio
  - Dublin Methodist Hospital, Dublin, Ohio
  - Mercy Cancer Center-Elyria, Elyria, Ohio
  - Armes Family Cancer Center, Findlay, Ohio
  - Blanchard Valley Hospital, Findlay, Ohio
  - Orion Cancer Care, Findlay, Ohio
  - Atrium Medical Center-Middletown Regional Hospital, Franklin, Ohio
  - Dayton Physicians LLC-Atrium, Franklin, Ohio
  - Central Ohio Breast and Endocrine Surgery, Gahanna, Ohio
  - Dayton Physicians LLC-Wayne, Greenville, Ohio
  - Wayne Hospital, Greenville, Ohio
  - Mount Carmel Grove City Hospital, Grove City, Ohio
  - Greater Dayton Cancer Center, Kettering, Ohio
  - First Dayton Cancer Care, Kettering, Ohio
  - Kettering Medical Center, Kettering, Ohio
  - Fairfield Medical Center, Lancaster, Ohio
  - OhioHealth Mansfield Hospital, Mansfield, Ohio
  - Marietta Memorial Hospital, Marietta, Ohio
  - OhioHealth Marion General Hospital, Marion, Ohio
  - UH Seidman Cancer Center at Landerbrook Health Center, Mayfield Heights, Ohio
  - UH Seidman Cancer Center at Lake Health Mentor Campus, Mentor, Ohio
  - UH Seidman Cancer Center at Southwest General Hospital, Middleburg Heights, Ohio
  - Knox Community Hospital, Mount Vernon, Ohio
  - Licking Memorial Hospital, Newark, Ohio
  - Newark Radiation Oncology, Newark, Ohio
  - University Hospitals Parma Medical Center, Parma, Ohio
  - Southern Ohio Medical Center, Portsmouth, Ohio
  - University Hospitals Portage Medical Center, Ravenna, Ohio
  - UH Seidman Cancer Center at Firelands Regional Medical Center, Sandusky, Ohio
  - Springfield Regional Cancer Center, Springfield, Ohio
  - Springfield Regional Medical Center, Springfield, Ohio
  - Dayton Physicians LLC-Upper Valley, Troy, Ohio
  - Upper Valley Medical Center, Troy, Ohio
  - University Hospitals Sharon Health Center, Wadsworth, Ohio
  - Saint Joseph Warren Hospital, Warren, Ohio
  - University Pointe, West Chester, Ohio
  - Saint Ann's Hospital, Westerville, Ohio
  - UH Seidman Cancer Center at Saint John Medical Center, Westlake, Ohio
  - UHHS-Westlake Medical Center, Westlake, Ohio
  - Saint Elizabeth Youngstown Hospital, Youngstown, Ohio
  - Genesis Healthcare System Cancer Care Center, Zanesville, Ohio
  - Cancer Centers of Southwest Oklahoma Research, Lawton, Oklahoma
  - University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma
  - Mercy Hospital Oklahoma City, Oklahoma City, Oklahoma
  - Cancer Treatment Centers of America, Tulsa, Oklahoma
  - Oklahoma Cancer Specialists and Research Institute-Tulsa, Tulsa, Oklahoma
  - Saint Alphonsus Medical Center-Baker City, Baker City, Oregon
  - Saint Charles Health System, Bend, Oregon
  - Clackamas Radiation Oncology Center, Clackamas, Oregon
  - Providence Cancer Institute Clackamas Clinic, Clackamas, Oregon
  - Bay Area Hospital, Coos Bay, Oregon
  - Good Samaritan Hospital, Corvallis, Oregon
  - Legacy Mount Hood Medical Center, Gresham, Oregon
  - Providence Newberg Medical Center, Newberg, Oregon
  - Saint Alphonsus Medical Center-Ontario, Ontario, Oregon
  - Legacy Good Samaritan Hospital and Medical Center, Portland, Oregon
  - Providence Portland Medical Center, Portland, Oregon
  - Providence Saint Vincent Medical Center, Portland, Oregon
  - Oregon Health and Science University, Portland, Oregon
  - Saint Charles Health System-Redmond, Redmond, Oregon
  - Legacy Meridian Park Hospital, Tualatin, Oregon
  - Christiana Care Health System-Concord Health Center, Chadds Ford, Pennsylvania
  - Thomas Jefferson University Hospital, Philadelphia, Pennsylvania
  - Eastern Regional Medical Center, Philadelphia, Pennsylvania
  - AnMed Health Cancer Center, Anderson, South Carolina
  - Prisma Health Cancer Institute - Spartanburg, Boiling Springs, South Carolina
  - Prisma Health Cancer Institute - Easley, Easley, South Carolina
  - Gibbs Cancer Center-Gaffney, Gaffney, South Carolina
  - Saint Francis Hospital, Greenville, South Carolina
  - Prisma Health Cancer Institute - Butternut, Greenville, South Carolina
  - Prisma Health Cancer Institute - Faris, Greenville, South Carolina
  - Prisma Health Greenville Memorial Hospital, Greenville, South Carolina
  - Saint Francis Cancer Center, Greenville, South Carolina
  - Prisma Health Cancer Institute - Eastside, Greenville, South Carolina
  - Prisma Health Cancer Institute - Greer, Greer, South Carolina
  - Gibbs Cancer Center-Pelham, Greer, South Carolina
  - Prisma Health Cancer Institute - Seneca, Seneca, South Carolina
  - Spartanburg Medical Center, Spartanburg, South Carolina
  - MGC Hematology Oncology-Union, Union, South Carolina
  - Sanford Cancer Center Oncology Clinic, Sioux Falls, South Dakota
  - Sanford USD Medical Center - Sioux Falls, Sioux Falls, South Dakota
  - Wellmont Bristol Regional Medical Center, Bristol, Tennessee
  - Memorial Hospital, Chattanooga, Tennessee
  - Baptist Memorial Hospital and Cancer Center-Collierville, Collierville, Tennessee
  - Cookeville Regional Medical Center, Cookeville, Tennessee
  - Vanderbilt-Ingram Cancer Center at Franklin, Franklin, Tennessee
  - Vanderbilt-Ingram Cancer Center Cool Springs, Franklin, Tennessee
  - The West Clinic - Wolf River, Germantown, Tennessee
  - Pulmonary Medicine Center of Chattanooga-Hixson, Hixson, Tennessee
  - Regional Cancer Center at Indian Path Community Hospital, Kingsport, Tennessee
  - Wellmont Holston Valley Hospital and Medical Center, Kingsport, Tennessee
  - The West Clinic - Mid-Town, Memphis, Tennessee
  - Baptist Memorial Hospital and Cancer Center-Memphis, Memphis, Tennessee
  - Vanderbilt Breast Center at One Hundred Oaks, Nashville, Tennessee
  - Vanderbilt University/Ingram Cancer Center, Nashville, Tennessee
  - Memorial GYN Plus, Ooltewah, Tennessee
  - Hendrick Medical Center, Abilene, Texas
  - Saint Joseph Regional Cancer Center, Bryan, Texas
  - Parkland Memorial Hospital, Dallas, Texas
  - UT Southwestern/Simmons Cancer Center-Dallas, Dallas, Texas
  - UT Southwestern/Simmons Cancer Center-Fort Worth, Fort Worth, Texas
  - Baylor College of Medicine/Dan L Duncan Comprehensive Cancer Center, Houston, Texas
  - Ben Taub General Hospital, Houston, Texas
  - M D Anderson Cancer Center, Houston, Texas
  - Michael E DeBakey VA Medical Center, Houston, Texas
  - UT Southwestern Clinical Center at Richardson/Plano, Richardson, Texas
  - University of Texas Health Science Center at San Antonio, San Antonio, Texas
  - Farmington Health Center, Farmington, Utah
  - University of Utah Sugarhouse Health Center, Salt Lake City, Utah
  - Huntsman Cancer Institute/University of Utah, Salt Lake City, Utah
  - Central Vermont Medical Center/National Life Cancer Treatment, Berlin Corners, Vermont
  - University of Vermont Medical Center, Burlington, Vermont
  - University of Vermont and State Agricultural College, Burlington, Vermont
  - Wellmont Medical Associates-Bristol, Bristol, Virginia
  - Southwest VA Regional Cancer Center, Norton, Virginia
  - VCU Massey Cancer Center at Stony Point, Richmond, Virginia
  - Virginia Commonwealth University/Massey Cancer Center, Richmond, Virginia
  - Providence Regional Cancer System-Aberdeen, Aberdeen, Washington
  - Overlake Medical Center, Bellevue, Washington
  - PeaceHealth Saint Joseph Medical Center, Bellingham, Washington
  - Harrison HealthPartners Hematology and Oncology-Bremerton, Bremerton, Washington
  - Harrison Medical Center, Bremerton, Washington
  - Highline Medical Center-Main Campus, Burien, Washington
  - Providence Regional Cancer System-Centralia, Centralia, Washington
  - Swedish Cancer Institute-Edmonds, Edmonds, Washington
  - Saint Elizabeth Hospital, Enumclaw, Washington
  - Providence Regional Cancer Partnership, Everett, Washington
  - Saint Francis Hospital, Federal Way, Washington
  - Swedish Cancer Institute-Issaquah, Issaquah, Washington
  - Kadlec Clinic Hematology and Oncology, Kennewick, Washington
  - Providence Regional Cancer System-Lacey, Lacey, Washington
  - Saint Clare Hospital, Lakewood, Washington
  - PeaceHealth Saint John Medical Center, Longview, Washington
  - Harrison HealthPartners Hematology and Oncology-Poulsbo, Poulsbo, Washington
  - Valley Medical Center, Renton, Washington
  - Pacific Gynecology Specialists, Seattle, Washington
  - Swedish Medical Center-Ballard Campus, Seattle, Washington
  - Kaiser Permanente Washington, Seattle, Washington
  - Swedish Medical Center-First Hill, Seattle, Washington
  - Swedish Medical Center-Cherry Hill, Seattle, Washington
  - PeaceHealth United General Medical Center, Sedro-Woolley, Washington
  - Providence Regional Cancer System-Shelton, Shelton, Washington
  - Franciscan Research Center-Northwest Medical Plaza, Tacoma, Washington
  - Northwest Medical Specialties PLLC, Tacoma, Washington
  - PeaceHealth Southwest Medical Center, Vancouver, Washington
  - Legacy Cancer Institute Medical Oncology and Day Treatment, Vancouver, Washington
  - Legacy Salmon Creek Hospital, Vancouver, Washington
  - Providence Saint Mary Regional Cancer Center, Walla Walla, Washington
  - Providence Regional Cancer System-Yelm, Yelm, Washington
  - United Hospital Center, Bridgeport, West Virginia
  - WVUH-Berkely Medical Center, Martinsburg, West Virginia
  - West Virginia University Healthcare, Morgantown, West Virginia
  - Camden Clark Medical Center, Parkersburg, West Virginia
  - Duluth Clinic Ashland, Ashland, Wisconsin
  - Northwest Wisconsin Cancer Center, Ashland, Wisconsin
  - Aurora Cancer Care-Southern Lakes VLCC, Burlington, Wisconsin
  - Marshfield Clinic-Chippewa Center, Chippewa Falls, Wisconsin
  - Marshfield Medical Center-EC Cancer Center, Eau Claire, Wisconsin
  - Mayo Clinic Health System-Eau Claire Clinic, Eau Claire, Wisconsin
  - Aurora Health Center-Fond du Lac, Fond du Lac, Wisconsin
  - Aurora Health Care Germantown Health Center, Germantown, Wisconsin
  - Aurora Cancer Care-Grafton, Grafton, Wisconsin
  - Bellin Memorial Hospital, Green Bay, Wisconsin
  - Saint Vincent Hospital Cancer Center Green Bay, Green Bay, Wisconsin
  - Saint Vincent Hospital Cancer Center at Saint Mary's, Green Bay, Wisconsin
  - Aurora BayCare Medical Center, Green Bay, Wisconsin
  - Aurora Cancer Care-Kenosha South, Kenosha, Wisconsin
  - Gundersen Lutheran Medical Center, La Crosse, Wisconsin
  - Mayo Clinic Health System-Franciscan Healthcare, La Crosse, Wisconsin
  - Marshfield Clinic - Ladysmith Center, Ladysmith, Wisconsin
  - University of Wisconsin Hospital and Clinics, Madison, Wisconsin
  - Aurora Bay Area Medical Group-Marinette, Marinette, Wisconsin
  - Marshfield Medical Center-Marshfield, Marshfield, Wisconsin
  - Aurora Cancer Care-Milwaukee, Milwaukee, Wisconsin
  - Aurora Saint Luke's Medical Center, Milwaukee, Wisconsin
  - Aurora Sinai Medical Center, Milwaukee, Wisconsin
  - Marshfield Clinic-Minocqua Center, Minocqua, Wisconsin
  - ProHealth D N Greenwald Center, Mukwonago, Wisconsin
  - Cancer Center of Western Wisconsin, New Richmond, Wisconsin
  - ProHealth Oconomowoc Memorial Hospital, Oconomowoc, Wisconsin
  - Saint Vincent Hospital Cancer Center at Oconto Falls, Oconto Falls, Wisconsin
  - Vince Lombardi Cancer Clinic - Oshkosh, Oshkosh, Wisconsin
  - Aurora Cancer Care-Racine, Racine, Wisconsin
  - Marshfield Medical Center-Rice Lake, Rice Lake, Wisconsin
  - Vince Lombardi Cancer Clinic-Sheboygan, Sheboygan, Wisconsin
  - Marshfield Clinic Stevens Point Center, Stevens Point, Wisconsin
  - Saint Vincent Hospital Cancer Center at Sturgeon Bay, Sturgeon Bay, Wisconsin
  - Aurora Medical Center in Summit, Summit, Wisconsin
  - Vince Lombardi Cancer Clinic-Two Rivers, Two Rivers, Wisconsin
  - ProHealth Waukesha Memorial Hospital, Waukesha, Wisconsin
  - UW Cancer Center at ProHealth Care, Waukesha, Wisconsin
  - Marshfield Clinic-Wausau Center, Wausau, Wisconsin
  - Aurora Cancer Care-Milwaukee West, Wauwatosa, Wisconsin
  - Aurora West Allis Medical Center, West Allis, Wisconsin
  - Marshfield Clinic - Weston Center, Weston, Wisconsin
  - Marshfield Clinic - Wisconsin Rapids Center, Wisconsin Rapids, Wisconsin
  - Billings Clinic-Cody, Cody, Wyoming
  - Welch Cancer Center, Sheridan, Wyoming

REFERENCES:
- [Derived] Shroff RT, King G, Colby S, Scott AJ, Borad MJ, Goff L, Matin K, Mahipal A, Kalyan A, Javle MM, El Dika I, Tan B, Cheema P, Patel A, Iyer R, Kelley RK, Thumar J, El-Khoueiry A, Guthrie KA, Chiorean EG, Hochster H, Philip PA. SWOG S1815: A Phase III Randomized Trial of Gemcitabine, Cisplatin, and Nab-Paclitaxel Versus Gemcitabine and Cisplatin in Newly Diagnosed, Advanced Biliary Tract Cancers. J Clin Oncol. 2025 Feb 10;43(5):536-544. doi: 10.1200/JCO-24-01383. Epub 2024 Dec 13. PMID 39671534

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 452 participants were registered to the study, 10 were ineligible and 1 was not analyzable.
Groups:
- Gem+Cisplatin+Nab-paclitaxel: Patients receive nab-paclitaxel IV over 30 minutes, cisplatin IV over 60 minutes, and gemcitabine hydrochloride IV over 30 minutes on days 1 and 8. Courses repeat every 21 days in the absence of disease progression or unacceptable toxicity.
- Gemcitabine + Cisplatin: Patients receive cisplatin IV over 60 minutes and gemcitabine hydrochloride IV over 30 minutes on days 1 and 8. Courses repeat every 21 days in the absence of disease progression or unacceptable toxicity.
Period: Overall Study
Arm/Group | Gem+Cisplatin+Nab-paclitaxel | Gemcitabine + Cisplatin
Started | 294 | 147
Completed | 0 | 0
Not Completed | 294 | 147
Not completed — Adverse Event or side effects | 72 | 28
Not completed — Refusal unrelated to adverse event | 33 | 33
Not completed — Progression/relapse | 132 | 60
Not completed — Death | 9 | 6
Not completed — Other - not protocol specified | 45 | 18
Not completed — Reason under review | 3 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Gem+Cisplatin+Nab-paclitaxel | Gemcitabine + Cisplatin | Total
Number analyzed (Participants) | 294 | 147 | 441
Age, Continuous [Median (Full Range); unit: years] | 63.2 [23.2 to 88.8] | 63.9 [23.2 to 83.6] | 63.5 [23.2 to 88.8]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 162 | 81 | 243
  Male | 132 | 66 | 198
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 30 | 15 | 45
  Not Hispanic or Latino | 256 | 125 | 381
  Unknown or Not Reported | 8 | 7 | 15
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 2 | 1 | 3
  Asian | 14 | 7 | 21
  Native Hawaiian or Other Pacific Islander | 1 | 0 | 1
  Black or African American | 18 | 7 | 25
  White | 244 | 119 | 363
  More than one race | 0 | 1 | 1
  Unknown or Not Reported | 15 | 12 | 27
Disease Site [Count of Participants; unit: Participants]
  Gallbladder adenocarcinoma | 46 | 24 | 70
  Intrahepatic cholangiocarcinoma | 198 | 99 | 297
  Extrahepatic cholangiocarcinoma | 50 | 24 | 74
Disease Stage [Count of Participants; unit: Participants]
  Locally advances | 77 | 41 | 118
  Metastatic | 217 | 106 | 323
Performance Status [Count of Participants; unit: Participants] — Zubrod Performance Status Scale range from 0 to 1, with higher scores reflecting greater disability.
  0: Fully active, able to carry on all pre-disease performance without restriction.
  1: Restricted in physically strenuous activity but ambulatory and able to carry out work of a light or sedentary nature, e.g., light housework, office work.
  Participants
    0 | 147 | 75 | 222
    1 | 147 | 72 | 219

OUTCOME MEASURES:

1. Primary Outcome: Overall Survival (OS)
Description: OS will be determined using the log-rank test with stratification by disease site (gallbladder adenocarcinoma versus [vs.] intrahepatic cholangiocarcinoma vs. extrahepatic cholangiocarcinoma), disease stage (locally advanced vs. metastatic), and Zubrod performance status (0 vs. 1). Distributions of overall survival by treatment arm will be estimated using the method of Kaplan-Meier.
Time Frame: Up to 3 years
Population: This population includes the 441 eligible and evaluable participants. 294 in the Gem+Cisplatin+Nab-paclitaxel arm and 147 in the Gemcitabine + Cisplatin arm.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Gem+Cisplatin+Nab-paclitaxel | Gemcitabine + Cisplatin
Number analyzed (Participants) | 294 | 147
months | 14.0 [12.4 to 16.1] | 13.6 [9.7 to 16.6]
Statistical Analysis 1: Comparison: Gem+Cisplatin+Nab-paclitaxel vs Gemcitabine + Cisplatin; Test type: Superiority; p = 0.41, Log Rank; Hazard Ratio (HR) = 0.91, 95% CI 2-sided [0.72 to 1.14]

2. Secondary Outcome: Number of Participants With Gr 3 Through 5 Adverse Events That Are Related to Study Drugs.
Description: Only adverse events that are possibly, probably, or definitely related to study drugs are reported. CTCAE Version 5.0 was used for all AE reporting.
Time Frame: Duration of treatment and follow-up until death or 3 years post registration.
Population: Participants who were eligible and received at least one dose of protocol treatment.
Measure: Number; unit: Participants
Arm/Group | Gem+Cisplatin+Nab-paclitaxel | Gemcitabine + Cisplatin
Number analyzed (Participants) | 287 | 134
Participants
  Abdominal pain | 2 | 0
  Acute kidney injury | 5 | 3
  Alanine aminotransferase increased | 6 | 1
  Alkaline phosphatase increased | 3 | 1
  Anemia | 95 | 30
  Anorexia | 8 | 0
  Arthralgia | 1 | 0
  Ascites | 2 | 0
  Aspartate aminotransferase increased | 5 | 0
  Ataxia | 1 | 0
  Atrial fibrillation | 1 | 0
  Back pain | 1 | 0
  Blood and lymphatic system disorders - Other, spec | 1 | 1
  Blood bilirubin increased | 3 | 1
  Cardiac arrest | 1 | 0
  Catheter related infection | 0 | 1
  Cholecystitis | 1 | 0
  Chronic kidney disease | 2 | 1
  Colitis | 2 | 0
  Constipation | 1 | 0
  Creatinine increased | 1 | 0
  Death NOS | 1 | 1
  Dehydration | 4 | 2
  Delirium | 1 | 0
  Diarrhea | 13 | 1
  Dizziness | 1 | 0
  Dysphagia | 1 | 0
  Dyspnea | 0 | 2
  Edema limbs | 4 | 0
  Endocarditis infective | 0 | 1
  Enterocolitis | 1 | 0
  Enterocolitis infectious | 3 | 0
  Epistaxis | 2 | 0
  Esophagitis | 1 | 0
  Fatigue | 27 | 8
  Febrile neutropenia | 10 | 2
  Fever | 1 | 0
  Flu like symptoms | 2 | 0
  GGT increased | 2 | 0
  Gallbladder infection | 0 | 1
  Gastric hemorrhage | 1 | 0
  Gastrointestinal disorders - Other, specify | 1 | 0
  General disorders and administration site conditio | 1 | 0
  Generalized muscle weakness | 3 | 1
  Headache | 1 | 0
  Hearing impaired | 1 | 0
  Heart failure | 0 | 1
  Hematuria | 1 | 0
  Hepatic infection | 1 | 1
  Hepatobiliary disorders - Other, specify | 2 | 0
  Hyperglycemia | 0 | 1
  Hyperkalemia | 2 | 0
  Hypertension | 7 | 1
  Hypoalbuminemia | 5 | 1
  Hypocalcemia | 3 | 1
  Hypokalemia | 9 | 2
  Hypomagnesemia | 6 | 5
  Hyponatremia | 6 | 4
  Hypotension | 3 | 1
  Infections and infestations - Other, specify | 3 | 2
  Infusion related reaction | 0 | 1
  Investigations - Other, specify | 1 | 0
  Lung infection | 2 | 0
  Lymphocyte count decreased | 30 | 4
  Memory impairment | 1 | 0
  Mucositis oral | 2 | 0
  Multi-organ failure | 1 | 0
  Muscle weakness lower limb | 1 | 0
  Myalgia | 1 | 0
  Nausea | 11 | 1
  Neutrophil count decreased | 105 | 37
  Pain | 1 | 0
  Paresthesia | 1 | 0
  Peripheral motor neuropathy | 1 | 0
  Peripheral sensory neuropathy | 10 | 1
  Peritoneal infection | 0 | 1
  Platelet count decreased | 56 | 20
  Pleural effusion | 1 | 0
  Portal vein thrombosis | 0 | 1
  Rectal hemorrhage | 1 | 0
  Respiratory failure | 1 | 0
  Respiratory, thoracic and mediastinal disorders - | 1 | 0
  Seizure | 0 | 1
  Sepsis | 15 | 3
  Skin infection | 4 | 1
  Superior vena cava syndrome | 1 | 0
  Supraventricular tachycardia | 1 | 0
  Syncope | 2 | 1
  Thromboembolic event | 9 | 1
  Thrush | 1 | 0
  Typhlitis | 1 | 0
  Upper gastrointestinal hemorrhage | 2 | 0
  Urinary tract infection | 4 | 1
  Vascular access complication | 1 | 0
  Vasovagal reaction | 1 | 0
  Vomiting | 5 | 0
  Wheezing | 0 | 1
  White blood cell decreased | 46 | 10

3. Secondary Outcome: Progression-free Survival (PFS)
Description: Distributions of PFS will be described using cumulative incidence estimates with differences in these estimates between treatment arms assessed by a stratified Cox regression model.
Time Frame: From date of registration to date of first documentation of progression or symptomatic deterioration, or death due to any cause, assessed up to 3 years
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Gem+Cisplatin+Nab-paclitaxel | Gemcitabine + Cisplatin
Number analyzed (Participants) | 294 | 147
months | 7.5 [6.4 to 8.5] | 6.3 [4.4 to 8.2]

4. Secondary Outcome: Overall Response Rate (ORR) as Measured by Response Evaluation Criteria in Solid Tumors (RECIST) 1.1 Criteria
Description: ORR is defined as confirmed and unconfirmed; complete response + partial response + stable disease. The chi-square test will be used to compare ORR, disease control rate (DCR), and rates of toxicity events across arms. ORR will be assessed in the subset of patients with measurable disease.
Time Frame: Up to 3 years
Measure: Count of Participants; unit: Participants
Arm/Group | Gem+Cisplatin+Nab-paclitaxel | Gemcitabine + Cisplatin
Number analyzed (Participants) | 290 | 146
Participants
  Complete Response | 6 | 1
  Partial Response | 55 | 11
  Unconfirmed Partial Response | 30 | 19
  Stable/No Response | 134 | 67
  Increasing Disease | 38 | 22
  Symptomatic Deterioration | 2 | 3
  Assessment Inadaquate | 25 | 23

5. Secondary Outcome: Disease Control Rate as Measured by RECIST 1.1 Criteria
Description: The chi-square test will be used to compare ORR, DCR, and rates of toxicity events across arms. Disease control includes confirmed and unconfirmed complete response, confirmed and unconfirmed partial response, and stable disease. In patients with non-measurable disease, disease control will be defined as those who are alive without disease progression.
Time Frame: Up to 3 years
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Gem+Cisplatin+Nab-paclitaxel | Gemcitabine + Cisplatin
Number analyzed (Participants) | 290 | 147
percentage of participants | 78 [72 to 82] | 67 [59 to 75]

6. Secondary Outcome: Changes in Carbohydrate Antigen 19-9 (CA 19-9) Levels
Description: Correlations between changes in CA19-9 levels from baseline to post-treatment and ORR will be estimated via logistic regression models, both within each treatment arm and in the overall cohort. Analyses will explore the prognostic and predictive values of CA19-9 for disease response.
Time Frame: Baseline up to course 3
Population: one participant had missing baseline CA and 96 participants had missing post-treatment CA. They were not included in the analysis
Measure: Median (Full Range); unit: U/mL
Arm/Group | Gem+Cisplatin+Nab-paclitaxel | Gemcitabine + Cisplatin
Number analyzed (Participants) | 237 | 102
U/mL | -12 [-151086 to 637797] | -2.97 [-283830 to 3318]

ADVERSE EVENTS:
Time Frame: Duration of treatment and follow up until death or 3 years post registration.
Groups:
- Gem+Cisplatin+Nab-paclitaxel: Patients receive nab-paclitaxel IV over 30 minutes, cisplatin IV over 60 minutes, and gemcitabine hydrochloride IV over 30 minutes on days 1 and 8. Courses repeat every 21 days in the absence of disease progression or unacceptable toxicity. The number of participants at risk in All-cause Mortality are the number of participants included in the primary analysis.
- Gemcitabine + Cisplatin: Patients receive cisplatin IV over 60 minutes and gemcitabine hydrochloride IV over 30 minutes on days 1 and 8. Courses repeat every 21 days in the absence of disease progression or unacceptable toxicity. The number of participants at risk in All-cause Mortality are the number of participants included in the primary analysis.
Arm/Group | Gem+Cisplatin+Nab-paclitaxel | Gemcitabine + Cisplatin
All-Cause Mortality (participants affected / at risk) | 237/294 | 115/147
Serious Adverse Events (participants affected / at risk) | 27/287 | 11/134
Other Adverse Events (participants affected / at risk) | 280/287 | 133/134
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Gem+Cisplatin+Nab-paclitaxel (N=287) | Gemcitabine + Cisplatin (N=134)
Anemia (Blood and lymphatic system disorders) | 2 | 0
Febrile neutropenia (Blood and lymphatic system disorders) | 3 | 0
Cardiac arrest (Cardiac disorders) | 1 | 0
Myocardial infarction (Cardiac disorders) | 1 | 0
Abdominal distension (Gastrointestinal disorders) | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 3 | 0
Enterocolitis (Gastrointestinal disorders) | 1 | 0
Gastric hemorrhage (Gastrointestinal disorders) | 1 | 0
Nausea (Gastrointestinal disorders) | 1 | 0
Small intestinal obstruction (Gastrointestinal disorders) | 2 | 0
Upper gastrointestinal hemorrhage (Gastrointestinal disorders) | 2 | 0
Death NOS (General disorders) | 1 | 2
Disease progression (General disorders) | 2 | 0
Fatigue (General disorders) | 2 | 0
Multi-organ failure (General disorders) | 1 | 0
Portal vein thrombosis (Hepatobiliary disorders) | 1 | 0
Biliary tract infection (Infections and infestations) | 2 | 0
Infections and infestations-Other (Infections and infestations) | 1 | 1
Sepsis (Infections and infestations) | 6 | 4
Alanine aminotransferase increased (Investigations) | 1 | 0
Alkaline phosphatase increased (Investigations) | 1 | 0
Aspartate aminotransferase increased (Investigations) | 1 | 0
Neutrophil count decreased (Investigations) | 3 | 0
Platelet count decreased (Investigations) | 3 | 2
White blood cell decreased (Investigations) | 1 | 0
Dehydration (Metabolism and nutrition disorders) | 1 | 0
Hypoglycemia (Metabolism and nutrition disorders) | 0 | 1
Hypokalemia (Metabolism and nutrition disorders) | 1 | 0
Hyponatremia (Metabolism and nutrition disorders) | 1 | 0
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 1 | 0
Neoplasms benign, malignant and unspecified (incl (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 2
Stroke (Nervous system disorders) | 1 | 0
Syncope (Nervous system disorders) | 0 | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 2 | 1
Respiratory, thoracic and mediastinal disorders-Ot (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Surgical and medical procedures-Other (Surgical and medical procedures) | 1 | 0
Hypotension (Vascular disorders) | 1 | 1
Superior vena cava syndrome (Vascular disorders) | 1 | 0
Thromboembolic event (Vascular disorders) | 2 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Gem+Cisplatin+Nab-paclitaxel (N=287) | Gemcitabine + Cisplatin (N=134)
Anemia (Blood and lymphatic system disorders) | 236 | 85
Blood and lymphatic system disorders-Other (Blood and lymphatic system disorders) | 15 | 4
Sinus tachycardia (Cardiac disorders) | 31 | 17
Tinnitus (Ear and labyrinth disorders) | 26 | 15
Blurred vision (Eye disorders) | 21 | 6
Eye disorders-Other (Eye disorders) | 17 | 4
Abdominal distension (Gastrointestinal disorders) | 20 | 8
Abdominal pain (Gastrointestinal disorders) | 105 | 51
Ascites (Gastrointestinal disorders) | 21 | 9
Bloating (Gastrointestinal disorders) | 17 | 9
Constipation (Gastrointestinal disorders) | 153 | 72
Diarrhea (Gastrointestinal disorders) | 138 | 47
Dry mouth (Gastrointestinal disorders) | 16 | 4
Dyspepsia (Gastrointestinal disorders) | 26 | 11
Dysphagia (Gastrointestinal disorders) | 15 | 3
Gastroesophageal reflux disease (Gastrointestinal disorders) | 38 | 13
Gastrointestinal disorders-Other (Gastrointestinal disorders) | 22 | 9
Mucositis oral (Gastrointestinal disorders) | 35 | 15
Nausea (Gastrointestinal disorders) | 176 | 88
Vomiting (Gastrointestinal disorders) | 87 | 46
Chills (General disorders) | 37 | 18
Edema face (General disorders) | 8 | 7
Edema limbs (General disorders) | 106 | 41
Fatigue (General disorders) | 222 | 99
Fever (General disorders) | 74 | 23
Flu like symptoms (General disorders) | 22 | 4
General disorders and administration site conditio (General disorders) | 20 | 5
Generalized edema (General disorders) | 20 | 6
Localized edema (General disorders) | 4 | 8
Non-cardiac chest pain (General disorders) | 18 | 5
Pain (General disorders) | 42 | 28
Infections and infestations-Other (Infections and infestations) | 17 | 11
Sepsis (Infections and infestations) | 11 | 9
Skin infection (Infections and infestations) | 17 | 7
Thrush (Infections and infestations) | 22 | 2
Urinary tract infection (Infections and infestations) | 24 | 12
Bruising (Injury, poisoning and procedural complications) | 17 | 8
Fall (Injury, poisoning and procedural complications) | 18 | 4
Alanine aminotransferase increased (Investigations) | 105 | 37
Alkaline phosphatase increased (Investigations) | 90 | 45
Aspartate aminotransferase increased (Investigations) | 97 | 34
Blood bilirubin increased (Investigations) | 44 | 21
Creatinine increased (Investigations) | 60 | 30
Investigations-Other (Investigations) | 16 | 9
Lymphocyte count decreased (Investigations) | 87 | 28
Neutrophil count decreased (Investigations) | 168 | 77
Platelet count decreased (Investigations) | 167 | 52
Weight gain (Investigations) | 15 | 10
Weight loss (Investigations) | 57 | 16
White blood cell decreased (Investigations) | 121 | 47
Anorexia (Metabolism and nutrition disorders) | 114 | 45
Dehydration (Metabolism and nutrition disorders) | 42 | 15
Hypercalcemia (Metabolism and nutrition disorders) | 18 | 2
Hyperglycemia (Metabolism and nutrition disorders) | 69 | 33
Hyperkalemia (Metabolism and nutrition disorders) | 21 | 7
Hypoalbuminemia (Metabolism and nutrition disorders) | 97 | 33
Hypocalcemia (Metabolism and nutrition disorders) | 62 | 28
Hypokalemia (Metabolism and nutrition disorders) | 57 | 26
Hypomagnesemia (Metabolism and nutrition disorders) | 124 | 51
Hyponatremia (Metabolism and nutrition disorders) | 90 | 36
Arthralgia (Musculoskeletal and connective tissue disorders) | 28 | 16
Back pain (Musculoskeletal and connective tissue disorders) | 60 | 31
Bone pain (Musculoskeletal and connective tissue disorders) | 21 | 7
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 35 | 12
Myalgia (Musculoskeletal and connective tissue disorders) | 31 | 14
Pain in extremity (Musculoskeletal and connective tissue disorders) | 43 | 16
Dizziness (Nervous system disorders) | 86 | 28
Dysgeusia (Nervous system disorders) | 65 | 24
Headache (Nervous system disorders) | 74 | 37
Paresthesia (Nervous system disorders) | 18 | 11
Peripheral motor neuropathy (Nervous system disorders) | 25 | 6
Peripheral sensory neuropathy (Nervous system disorders) | 135 | 31
Anxiety (Psychiatric disorders) | 46 | 33
Depression (Psychiatric disorders) | 21 | 15
Insomnia (Psychiatric disorders) | 75 | 38
Chronic kidney disease (Renal and urinary disorders) | 11 | 7
Urinary frequency (Renal and urinary disorders) | 9 | 8
Cough (Respiratory, thoracic and mediastinal disorders) | 58 | 18
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 94 | 26
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 53 | 11
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 22 | 3
Rhinorrhea (Respiratory, thoracic and mediastinal disorders) | 15 | 4
Sore throat (Respiratory, thoracic and mediastinal disorders) | 16 | 7
Alopecia (Skin and subcutaneous tissue disorders) | 148 | 27
Dry skin (Skin and subcutaneous tissue disorders) | 16 | 7
Pruritus (Skin and subcutaneous tissue disorders) | 23 | 12
Rash acneiform (Skin and subcutaneous tissue disorders) | 20 | 5
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 53 | 14
Skin and subcutaneous tissue disorders-Other (Skin and subcutaneous tissue disorders) | 26 | 14
Hypertension (Vascular disorders) | 70 | 36
Hypotension (Vascular disorders) | 24 | 9
Thromboembolic event (Vascular disorders) | 44 | 18

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2021-06-13): https://cdn.clinicaltrials.gov/large-docs/14/NCT03768414/Prot_SAP_ICF_000.pdf